CLINICAL TRIAL: NCT07382661
Title: A Phase 1 Clinical Trial to Evaluate the Safety and the Pharmacokinetics Drug-drug Interaction of DW4421 and Amoxicillin/Clarithromycin in Healthy Adult Volunteers
Brief Title: Drug-Drug Interaction Between DW4421 and Amoxicillin/Clarithromycin
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DW4421-103
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Healthy Adult Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): A-B-C (A: DW4421 1T bid; B: DW4421-1 2C bid + DW4421-2 1T bid; C: DW4421 1T bid + DW4421-1 2C bid + DW4421-2 1T bid)
  Interventions: Drug: DW4421; Drug: DW4421-1; Drug: DW4421-2
- Sequence 2 (Experimental): A-C-B (A: DW4421 1T bid; B: DW4421-1 2C bid + DW4421-2 1T bid; C: DW4421 1T bid + DW4421-1 2C bid + DW4421-2 1T bid)
  Interventions: Drug: DW4421; Drug: DW4421-1; Drug: DW4421-2
- Sequence 3 (Experimental): B-A-B (A: DW4421 1T bid; B: DW4421-1 2C bid + DW4421-2 1T bid; C: DW4421 1T bid + DW4421-1 2C bid + DW4421-2 1T bid)
  Interventions: Drug: DW4421; Drug: DW4421-1; Drug: DW4421-2
- Sequence 4 (Experimental): B-C-A (A: DW4421 1T bid; B: DW4421-1 2C bid + DW4421-2 1T bid; C: DW4421 1T bid + DW4421-1 2C bid + DW4421-2 1T bid)
  Interventions: Drug: DW4421; Drug: DW4421-1; Drug: DW4421-2
- Sequence 5 (Experimental): C-A-B (A: DW4421 1T bid; B: DW4421-1 2C bid + DW4421-2 1T bid; C: DW4421 1T bid + DW4421-1 2C bid + DW4421-2 1T bid)
  Interventions: Drug: DW4421; Drug: DW4421-1; Drug: DW4421-2
- Sequence 6 (Experimental): C-B-A (A: DW4421 1T bid; B: DW4421-1 2C bid + DW4421-2 1T bid; C: DW4421 1T bid + DW4421-1 2C bid + DW4421-2 1T bid)
  Interventions: Drug: DW4421; Drug: DW4421-1; Drug: DW4421-2

INTERVENTIONS:
Drug: DW4421 — 1 tablet will be orally administered
Drug: DW4421-1 — 2 capsules will be orally administered
Drug: DW4421-2 — 1 tablet will be orally administered

SUMMARY:
Drug-Drug Interaction between DW4421 and Amoxicillin/Clarithromycin

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Healthy adult aged 19 to 50 (inclusive) years, at the time of screening.
* Subjects weighing between 50 kg and 90 kg with BMI between 18 and 27 kg/m2 (inclusive) at screening visit.

Exclusion Criteria:

* Those who have clinical significant liver, kidney, nervous system, respiratory, endocrine, hematology and oncology, cardiovascular, urinary, and mental diseases or past history.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Cmax,ss: Maximum concentration of DW4421, DW4421-1 and DW4421-2 at steady state | Up to day 6 or day 7
AUCτ,ss: Area under the drug concentration-time curve of DW4421, DW4421-1, DW4421-2 within a dosing interval at steady state | Up to day 6 or day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, North Chungcheong, South Korea